CLINICAL TRIAL: NCT06495905
Title: Evaluation of the Effectiveness and Safety of Transbronchoscopic Infusion of Amphotericin B + Inhalation of Amphotericin B + Transbronchoscopic Debridement + Systematic Antifungal Multimodal Treatment of Pulmonary Mucormycosis
Brief Title: Efficacy and Safety of Systematic Therapy and Bronchoscopic Interventional Treatment for Pulmonary Mucormycosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ST&BITPM
Record Dates: First submitted 2024-01-24; First posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-01

CONDITIONS: Pulmonary Mucormycosis
Keywords: pulmonary mucormycosis; bronchoscopy; treatment
MeSH Terms: interventions — liposomal amphotericin B; posaconazole; isavuconazole

STUDY DESIGN:
Intervention Model Description: Prospective, Intervention, observational, Propensity Matching Analysis study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Multimodal Treatment (Experimental): 1. combination drug therapy：liposomal amphotericin B + posaconazole or Isavuconazole：3-5mg/kg/day+ Posaconazole 300 mg once daily; target blood trough concentration is >1ug/mL; if posaconazole is unavailable, Isavuconazole 200 mg once daily may be an alternative.
  2. transbronchoscopic local precision infusion of amphotericin B: Maximum dose not more than 30mg per session
  3. transoral nebulized inhalation of amphotericin B：amphotericin B 10mg + 5ml of sterilized water for injection, inhalation 2/day.
  4)transbronchoscopic interventional debridement
  Interventions: Procedure: transbronchoscopic interventional debridement

INTERVENTIONS:
Procedure: transbronchoscopic interventional debridement — 1. combination drug therapy：liposomal amphotericin B + posaconazole or Isavuconazole：3-5mg/kg/day+ Posaconazole 300 mg once daily; target blood trough concentration is >1ug/mL; if posaconazole is unavailable, Isavuconazole 200 mg once daily may be an alternative.
  2. transbronchoscopic local precision infusion of amphotericin B: Maximum dose not more than 30mg per session
  3. transoral nebulized inhalation of amphotericin B：amphotericin B 10mg + 5ml of sterilized water for injection, inhalation 2/day.
  4)transbronchoscopic interventional debridement
  Other Names: transbronchoscopic local precision infusion of amphotericin B; transoral nebulized inhalation of amphotericin B; liposomal amphotericin B + posaconazole or Isavuconazole

SUMMARY:
Evaluation of the effectiveness and safety of transbronchoscopic local precision infusion of amphotericin B + transoral nebulized inhalation of amphotericin B + transbronchoscopic interventional debridement + liposomal amphotericin B + posaconazole or Isavuconazole multimodal treatment of pulmonary mucormycosis

DETAILED DESCRIPTION:
Key rationale for the treatment of mucormycosis is early surgical intervention, including local debridement and removal of infected tissues or organs if possible. Systemic antifungal therapy is also necessary for mucormycosis, including amphotericin B liposomes and deoxycholates, Isavuconazole, posaconazole, and so on. Antifungal drug therapy has a mortality rate of up to 40%, which can be reduced to 23% when combined with surgical treatment. However, some patients who are unable to tolerate surgical procedures on the chest when in bad condition, especially patients with hematological malignancies undergoing hematopoietic stem cell transplantation, are susceptible to multiple mucormycosis of the lungs, and the mortality rate of untreated systemically disseminated mucormycosis infections is high at 80%. Isavuconazole, so we aim to explore the multimodal treatment of liposomal amphotericin B + posaconazole or esaconazole + transbronchoscopic localized precise instillation of amphotericin B + oral nebulized inhalation of amphotericin B + transbronchoscopic interventional debridement to alleviate the pulmonary mucormycosis in chest imaging and reduce the mortality rate of patients with mucormycosis infection.

ELIGIBILITY:
Inclusion Criteria:

* Subjects suspected of pulmonary mucormycosis by clinical radiology will be enrolled in the study if the pathologic or microbiological diagnosis of mucormycosis (smear showing sterile mycelium, culture or molecular evidence of mucormycosis) is confirmed.
* Cases of diffuse mucormycosis will only be included if lung infection is confirmed pathologically or microbiologically by respiratory secretions or biopsy samples.
* Ability to tolerate bronchoscopy.

Exclusion Criteria:

* Pregnant and breastfeeding female patients
* Age <18 years
* Patients with HIV infection
* Contraindications to bronchoscopy (including platelet count < 100 x 109/L, active hemoptysis, severe respiratory or heart failure, severe arrhythmia, unstable angina or hypertension, severe pneumothorax or mediastinal emphysema, patients with acute myocardial infarction, cerebral infarction, and cerebral hemorrhage within 3 months
* Patients unable to tolerate bronchoscopy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-30 (Estimated); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
the rate of complete or partial response at 4 weeks | 4 weeks
  * Complete response: Resolution of all clinical signs and symptoms and more than 90% of lesions visible on radiology
  * Partial response: Clinical improvement and >50% improvement in findings on radiology

SECONDARY OUTCOMES:
the rate of complete or partial response at 12 weeks | 12 weeks
  * Complete response: Resolution of all clinical signs and symptoms and more than 90% of lesions visible on radiology
  * Partial response: Clinical improvement and >50% improvement in findings on radiology
Survival rate at 6 months | 6 months
  estimates using all-cause mortality at 12 months
the incidence of adverse reactions related to this comprehensive treatment at 4 weeks | 4 weeks
  The adverse reactions were assessed based on the Common Terminology Criteria for Adverse Events 5.0(CTCAE5.0)

CONTACTS AND LOCATIONS:
Overall Officials: Manting Liu, MD, Principal Investigator — Tsinghua University
Locations (1):
- Beijing TsingHua ChangGung hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Luo Q, He X, Xu J, Li L, Zhao L, Mu X. Reduced serum iron levels predict poor prognosis in pulmonary mucormycosis patients: a prospective, case-control study. Sci Rep. 2025 Aug 19;15(1):30395. doi: 10.1038/s41598-025-15186-3. PMID 40830172